CLINICAL TRIAL: NCT05178069
Title: Lactobacillus Rhamnosus GG: A Novel Probiotic Therapy for Treating Alcohol Use Disorder
Brief Title: LGG Supplementation in Patients With AUD and ALD
Acronym: AUD+ALD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Vatsalya Vatsalya, Faculty in Medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21.1038; K23AA029198 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2022-01-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder; Alcohol-associated Liver Disease
Keywords: AUD; ALD; AH; TLFB; LTDH; AUDIT; WHO Drinking Level Reduction Criteria; MELD; ALT; AST; ABIC; Total Bilirubin; Heavy Drinking; Drinking Pattern; AUD Domains; Albumin
MeSH Terms: conditions — Alcoholism | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Time by Treatment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator: Placebo for Probiotic (Placebo Comparator): Placebo capsule that matches the probiotic capsule in appearance will be given once daily for 180 days.
  Interventions: Drug: : Placebo for Probiotic
- Active Comparator: Lactobacillus Rhamnosus GG (Active Comparator): Dietary supplement capsule (Lactobacillus Rhamnosus GG) will be given once daily for 180 days.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus GG

INTERVENTIONS:
Drug: : Placebo for Probiotic — Capsule manufactured without active ingredients.
  Other Names: Dummy capsule
  Arms: Placebo Comparator: Placebo for Probiotic
Dietary Supplement: Lactobacillus Rhamnosus GG — Probiotic nutritional supplement; Lactobacillus Rhamnosus G
  Other Names: Culturelle
  Arms: Active Comparator: Lactobacillus Rhamnosus GG

SUMMARY:
To test the efficacy of 6-month LGG compared to placebo in treating Alcoholic Use Disorder (AUD) and liver injury in Alcoholic Hepatitis (AH). And to evaluate the effects of LGG treatment compared to placebo on therapeutic-mechanistic markers of the gut-brain axis and pro-inflammatory activity in patients with AUD and moderate AH

DETAILED DESCRIPTION:
Aim. 1: To test the efficacy of 6-month LGG compared to placebo in treating AUD: (1a) by lowering heavy drinking (1b) by reducing relapse episodes to minimal/absent incident level; (1c) by showing a significant positive effect on one or more of the underlying neurobehavioral domain, and (1d) by lowering a biochemical marker of alcohol intake.

Aim. 2: To test if 6-month LGG treatment compared to placebo will improve the symptoms and liver injury in AH: (2a) by significantly improving liver related tests (AST, ALT, AST:ALT, albumin, bilirubin and INR; K18M65 and K18M30) and clinical severity/prognostic markers (MELD, Maddrey); (2b) by substantially improving the overall health as assessed by the patient reported outcomes (Quality of Life [QOL] scale, and drinker inventory of consequences [DrInC]); and (2c) by lowering frequency and intensity of treatment/disease based adverse effects (AE).

Aim. 3: To evaluate the effects of LGG treatment compared to placebo on therapeutic-mechanistic markers of gut-brain axis and pro-inflammatory activity in patients with AUD and moderate AH: (3a) by identifying the blood biomarkers of gut-barrier dysfunction and endotoxemia, and inflammation; (3b) by determining the therapeutic targets of LGG involved in the gut-brain axis of AUD using LC-MS metabolomic fecal assays (candidate markers of gut-dysfunction associated neurotransmitters); and (3c) by validating the efficacy of LGG treatment vs. placebo to lower inflammation using an ex-vivo design.

ELIGIBILITY:
Inclusion Criteria:

1. Breath alcohol concentration (BAC) equal to 0.00 when the participant signs the informed consent document.
2. Age between 21 and 65 years old (inclusive).
3. Willingness to receive trial treatment.
4. Ability to provide informed consent
5. Understanding that this is not an alcohol treatment study.
6. Heavy drinking. Men must consume ≥ 20 and women ≥ 14 standardized alcoholic beverages a week for the past 3 months.
7. Diagnosis of Alcohol Use Disorder using DSM V criteria.
8. 50 <AST<400 U/L; AST > ALT; and ALT < 200 U/L; total bilirubin > 1.2 mg/dL
9. Model for End-Stage Liver Disease: 8 ≤ (MELD) ≤19.
10. Good health as confirmed by medical history, physical examination, ECG, laboratory tests and vital signs except for liver injury and AUD related history.
11. Provide contact information for someone who may be able to contact the subject in case of a missed appointment.
12. . Females of child-bearing potential must not be pregnant and must be using birth control

Exclusion Criteria:

1. Current (last 12 months) DSM V diagnosis of dependence on any psychoactive substance other than alcohol or nicotine,
2. Positive urine drug screen at baseline for any illegal substance other than marijuana,
3. History of hospitalization for alcohol intoxication delirium, alcohol withdrawal delirium or seizure,
4. Participation in any research study for alcoholism treatment within 3 months prior to signing the informed consent,
5. Pharmacological treatment with naltrexone, acamprosate, topiramate, or disulfiram within 1 month prior to randomization,
6. Lifetime diagnosis based on DSM-V criteria of schizophrenia, bipolar disorder, or other psychosis, eating disorders; current or past year diagnosis of major depression
7. In the investigators' opinion, moderate to severe risk of suicide (e.g., active plan, or recent attempt in last 6 months),
8. Current use of psychotropic medications that cannot be discontinued,
9. Clinically significant medical abnormalities (apart from moderate ALD, MELD≤19),
10. Clinical Institute Withdrawal Assessment for Alcohol revised (CIWA-Ar) >10, at screening for more than 3 days,
11. Serious medical diseases, such as cancer, liver cirrhosis, pancreatitis, severe alcohol associated hepatitis, heart chronic failure, chronic kidney failure, chronic intestinal diseases (e.g., Crohn's disease), chronic neurological disorders (e.g., tardive dyskinesia, epilepsy, Parkinson's disease)
12. History of clinically significant hypotension (e.g., history of lipotimia and/or syncopal episodes)
13. History of adverse reactions to needle puncture,
14. Obesity (BMI ≥ 33.0 kg/m2),
15. Pregnancy; incarceration; inability to provide consent
16. Signs of systemic infection: Fever > 38o C, positive blood or ascites cultures, on appropriate antibiotic therapy for > 3 days within 3 days of inclusion
17. Acute gastrointestinal bleeding requiring > 2 units blood transfusion within the previous 2 weeks
18. Undue risk from immunosuppression: Positive HBsAg; positive skin PPD skin test or history of treatment for tuberculosis; known HIV infection

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
By lowering heavy drinking to meet the criteria on the responder definitions of abstinence, no heavy drinking days, WHO 1-level, and WHO 2-level reduction | 180 days
  Timeline Followback for past 180 days [Unit: numerical frequency], AUDIT [Unit: numerical frequency], monthly drinking questionnaire [Unit: numerical frequency]).
By reducing relapse episodes to minimal/absent incident level | 180 days
  (Unit: incident frequency).
By showing a significant positive effect on one or more of the underlying neurobehavioral domains. | 180 days
  Questionnaires: reward (reasons for heavy drinking questionnaire or RHDQ [Unit: numerical frequency]), craving (Penn Alcohol Craving Scale or PACS, [Unit: numerical frequency]; and obsessive compulsive drinking scale or OCDS [Unit: numerical frequency]), withdrawal (Clinical Institute Withdrawal Assessment Alcohol Scale Revised [CIWA-AR] or CIWA-AR [Unit: numerical frequency]), and reinforcement effects (Desires for Alcohol Questionnaire or DAQ [Unit: numerical frequency]).
By lowering a biochemical marker of alcohol intake | 180 days
  PeTH (Unit: μmol/L)

SECONDARY OUTCOMES:
By significantly improving liver related and clinical markers | 180 days
  Liver markers: Aspartate transaminases or AST (Unit: IU/L), Alanine Transaminases or ALT (Unit: IU/L), Albumin (Unit: g/dL), Total bilirubin (Unit: mg/dL), Creatinine (Unit: mg/dL), and INR (Unit: numerical), AST:ALT ratio (numerical unit), Prothrombin Time or PT (Unit: seconds).
  Clinical marker: Model For End-Stage Liver Disease or MELD ([=0.957 × ln(Cr) + 0.378 × ln(bilirubin) + 1.120 × ln(INR) + 0.643]. Unit: numerical), Maddrey's Discriminant Function for Alcoholic Hepatitis or Maddrey DF ([=4.6 * (Pt's PT - Control PT) + TBili]. Unit: numerical).
  Laboratory markers: K18M65 and K18M30 (Unit for both: IU/L).
By substantially improving the overall health as assessed by the patient reported outcomes | 180 days
  Quality of Life or QOL scale [Unit: numerical frequency], Drinker inventory of consequences or DrInC [unit: numerical frequency].
By lowering frequency and intensity of treatment/disease based adverse effects (AE). | 180 days
  Incident frequency of AE [Unit: numerical], Severity Scale (AE/SAE (Unit: 1-5).

OTHER OUTCOMES:
To determine the therapeutic-mechanistic markers of gut-brain axis, pro-inflammatory activity in AUD | 180 days
  1. By identifying the blood biomarkers of gut-barrier dysfunction and endotoxemia as assessed by: LPS [Unit: EU/ml], LBP [Unit: ng/ml], sCD14 [Unit: x 10^6 pg/ml]. Serum Inflammation markers: IL1β, IL33, IL18, IL17, IL22, TNFα [Units for all: pg/ml].
  2. By determining the therapeutic targets of LGG involved in the gut-brain axis of AUD using LC-MS metabolomic fecal assays (candidate markers of gut-dysfunction associated neurotransmitters): Gamma Aminobutyric Acid or GABA [Unit: pmoles/ml], hexyl-2-methyl butyrate or HMBA (Unit: mmol/L), serotonin (Unit: ng/mL), dopamine (Unit: ng/ml), acetylcholine (Unit: nmol/L), tryptophan (Unit: umol/L), and short-chain fatty acids (Unit: mmol/L). Units can be relative in intensity (as fold-change).
  3. By validating the efficacy of LGG treatment vs. placebo to lower inflammation using an ex-vivo design: Candidate WBC type derived Inflammation markers: IL1β, IL33, IL18, IL17, IL22, TNFα [Units for all: pg/ml].

CONTACTS AND LOCATIONS:
Overall Officials: Vatsalya Vatsalya, MD, Principal Investigator — Department of Medicine, University of Louisville; Craig J McClain, MD, Study Chair — Department of Medicine, University of Louisville; Harsh Tiwari, MD, Study Director — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClain CJ, Vatsalya V, Mitchell MC. Keratin-18: Diagnostic, Prognostic, and Theragnostic for Alcohol-Associated Hepatitis. Am J Gastroenterol. 2021 Jan 1;116(1):77-79. doi: 10.14309/ajg.0000000000001042. PMID 33306505
- [Background] Gala KS, Vatsalya V. Emerging Noninvasive Biomarkers, and Medical Management Strategies for Alcoholic Hepatitis: Present Understanding and Scope. Cells. 2020 Feb 25;9(3):524. doi: 10.3390/cells9030524. PMID 32106390
- [Background] Vatsalya V, Cave MC, Kong M, Gobejishvili L, Falkner KC, Craycroft J, Mitchell M, Szabo G, McCullough A, Dasarathy S, Radaeva S, Barton B, McClain CJ. Keratin 18 Is a Diagnostic and Prognostic Factor for Acute Alcoholic Hepatitis. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2046-2054. doi: 10.1016/j.cgh.2019.11.050. Epub 2019 Dec 4. PMID 31811953
- [Background] Zhou Y, Vatsalya V, Gobejishvili L, Lamont RJ, McClain CJ, Feng W. Porphyromonas gingivalis as a Possible Risk Factor in the Development/Severity of Acute Alcoholic Hepatitis. Hepatol Commun. 2018 Dec 14;3(2):293-304. doi: 10.1002/hep4.1296. eCollection 2019 Feb. PMID 30766965
- [Background] Gowin JL, Sloan ME, Stangl BL, Vatsalya V, Ramchandani VA. Vulnerability for Alcohol Use Disorder and Rate of Alcohol Consumption. Am J Psychiatry. 2017 Nov 1;174(11):1094-1101. doi: 10.1176/appi.ajp.2017.16101180. Epub 2017 Aug 4. PMID 28774194
- [Background] Vatsalya V, Gowin JL, Schwandt ML, Momenan R, Coe MA, Cooke ME, Hommer DW, Bartlett S, Heilig M, Ramchandani VA. Effects of Varenicline on Neural Correlates of Alcohol Salience in Heavy Drinkers. Int J Neuropsychopharmacol. 2015 Jul 25;18(12):pyv068. doi: 10.1093/ijnp/pyv068. PMID 26209857
- [Background] Vatsalya V, Gala KS, Hassan AZ, Frimodig J, Kong M, Sinha N, Schwandt ML. Characterization of Early-Stage Alcoholic Liver Disease with Hyperhomocysteinemia and Gut Dysfunction and Associated Immune Response in Alcohol Use Disorder Patients. Biomedicines. 2020 Dec 24;9(1):7. doi: 10.3390/biomedicines9010007. PMID 33374263
- [Background] Vatsalya V, Kong M, Marsano LM, Kurlawala Z, Chandras KV, Schwandt ML, Ramchandani VA, McClain CJ. Interaction of Heavy Drinking Patterns and Depression Severity Predicts Efficacy of Quetiapine Fumarate XR in Lowering Alcohol Intake in Alcohol Use Disorder Patients. Subst Abuse. 2020 Sep 9;14:1178221820955185. doi: 10.1177/1178221820955185. eCollection 2020. PMID 32963470
- See also: Details of the Study at NIH Reporter — https://reporter.nih.gov/search/zmJAfR_IOkGNjlHYcbLx0w/project-details/10191836
- See also: Clinical Laboratory for the Intervention Development of AUD and Organ-Injury — https://louisville.edu/medicine/departments/medicine/divisions/gimedicine/faculty/vatsalya-lab